CLINICAL TRIAL: NCT00343902
Title: Randomized Clinical Trial of a Crataegus Oxycantha Extract in Chronic Heart Failure
Brief Title: Hawthorn Extract Randomized Blinded Chronic Heart Failure (HERB CHF) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P50AT000011 (NIH); 1999-0440
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2006-06-23 (Estimated); Status verified 2006-06

CONDITIONS: Chronic Heart Failure
Keywords: Hawthorn; Crataegus; Herbs

INTERVENTIONS:
Drug: Crataegus Special Extract WS 1442

SUMMARY:
To determine the effect of hawthorn extract 450 mg bid vs. placebo, in addition to standard medical therapy in ambulatory patients with NYHA class II to IV chronic heart failure on submaximal exercise as measured by the 6-minute walk test

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory individuals 18 years and older who had been diagnosed with CHF (NYHA functional classes II-IV) for > 3 months
* Left ventricular ejection fraction (LVEF) of ≤ 40 percent
* Receiving indicated standard therapy (if not contraindicated or intolerant for > 3 months) defined as a diuretic, an ACE-inhibitor or an angiotensin receptor blocker (ARB) and a beta-blocke
* Patients with NYHA class III or IV symptoms were also required to receive spironolactone. Doses of these drugs had to be stable for ≥ 3 months, except for diuretics, for which ≥ 1 month of stability was required.

Exclusion Criteria:

* Hemodynamically severe uncorrected primary valvular disease
* Active myocarditis
* Hypertrophic cardiomyopathy
* Restrictive cardiomyopathy
* Myocardial infarction, stroke, unstable angina, coronary artery bypass graft surgery, valvular surgery, or angioplasty < 3 months before randomization
* Symptomatic or sustained ventricular tachycardia not controlled by antiarrhythmic drugs or an implantable cardioverter-defibrillator
* Any condition other than heart failure that would be expected to limit exercise (e.g., angina, peripheral vascular disease, pulmonary disease, arthritis, or an orthopedic problem severe enough to limit exercise)
* Nursing mothers, pregnant women and those planning a pregnancy during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2000-01; Study Completion 2004-05

PRIMARY OUTCOMES:
Distance walked on a six minute walk test at six months

SECONDARY OUTCOMES:
Minnesota Living with Hearth Failure Questionnaire (Disease specific quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Aaronson, MD, MS, Principal Investigator — University of Michigan; Suzanna M Zick, ND, MPH, Principal Investigator — University of Michigan; Stephen Bolling, MD, Study Director — University of Michigan, Department of Surgery
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Zick SM, Blume A, Aaronson KD. The prevalence and pattern of complementary and alternative supplement use in individuals with chronic heart failure. J Card Fail. 2005 Oct;11(8):586-9. doi: 10.1016/j.cardfail.2005.06.427. PMID 16230260
- [Derived] Zick SM, Vautaw BM, Gillespie B, Aaronson KD. Hawthorn Extract Randomized Blinded Chronic Heart Failure (HERB CHF) trial. Eur J Heart Fail. 2009 Oct;11(10):990-9. doi: 10.1093/eurjhf/hfp116. PMID 19789403